CLINICAL TRIAL: NCT00679445
Title: A Feasibility Study to Evaluate the Safety And Tolerability of the EPI-RAD90™ Ophthalmic System for the Treatment of Subfoveal Choroidal Neovascularization (CNV) in Patients With Age-Related Macular Degeneration (AMD) That Have Failed Primary Anti-VEGF Therapy
Brief Title: A Study to Evaluate the Neovista Ophthalmic System for the Treatment of Subfoveal CNV in Patients With AMD That Have Failed Primary Anti-VEGF Therapy
Acronym: ROSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeoVista (Industry)
Responsible Party: Jeffrey Nau, MMS (Director, Clinical Affairs), NeoVista Incorporated
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVI-006
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: Macular; Degeneration; AMD; Wet Age-related macular degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Device: NeoVista Ophthalmic System A single procedure using the NeoVista Ophthalmic System plus an injection of Lucentis.
  Interventions: Device: NeoVista Ophthalmic System

INTERVENTIONS:
Device: NeoVista Ophthalmic System — A single procedure using the NeoVioasta Ophthalmic System plus an injection of Lucentis.

SUMMARY:
The objective of this clinical study is to evaluate the safety and feasibility of focal delivery of radiation for the treatment of subfoveal choroidal neovascularization (CNV) in patients with age related macular degeneration that have failed Primary Anti-VEGF therapy.

DETAILED DESCRIPTION:
Therapeutic advances in the arena of neovascular age-related macular degeneration (AMD) have provided multiple treatment options for the disease. Radiotherapy has been studied in multiple clinical trials in the past with many studies showing a therapeutic benefit. Treatment with radiotherapy and anti-VEGF compounds is a promising approach to treating AMD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have predominantly classic, minimally classic, or occult with no classic lesions, as determined by the Investigator, secondary to AMD, with a total lesion size (including blood, scarring, and neovascularization) of < 12 total disc areas (21.24 mm2), and a GLD ≤5.4 mm
* Subjects must have received a minimum of three (3) prior injections (a minimum of 3 prior injections of the same compound) of anti-VEGF therapy (Lucentis® or Avastin®, subjects may have been treated previously with Macugen®, but must have been most recently treated with Lucentis® or Avastin® and met the criteria for failure below) with evidence of "failure" to respond to therapy
* Subjects must be age 50 or older

Exclusion Criteria:

* Subjects with prior or subfoveal CNV therapy with photodynamic therapy, intravitreal or subretinal steroids, or transpupillary thermotherapy (TTT) (Note: This includes subjects with no known history, but with photographic evidence of prior therapy)
* Subjects who underwent previous radiation therapy to the eye, head or neck
* Subjects who have been previously diagnosed with Type 1 or Type 2 diabetes mellitus. Subjects who do not have a documented diagnosis but have retinal findings consistent with Type 1 or Type 2 Diabetes Mellitus.
* Women of child-bearing potential (female subjects must be post menopausal or surgically sterilized)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety Parameters to be evaluated include incidence and severity of ocular adverse events identified by eye examinations, including visual acuity. Retinal thickness will also be measured, and stereo fundus photography will be reviewed. | 3 Year

SECONDARY OUTCOMES:
Efficacy Assessment: Preliminary efficacy will be evaluated by measuring best-corrected visual acuity (ETDRS) and AMD lesion size and leakage as assessed by fluorescein angiography at 1, 2, 3, 6, 12, 18, 24, and 36 months in the study eye. | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Heier, MD, Principal Investigator — Ophthalmic Consultants of Boston; Jeffrey A Nau, MMS, Study Director — NeoVista, Inc; Michael Singer, MD, Principal Investigator — Medical Center Ophthalmology Associates
Locations (2):
- United States (2):
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Medical Center Ophthalmology Associates, San Antonio, Texas